CLINICAL TRIAL: NCT00321165
Title: The AOT (Acridine Orange and Taurolidine) Trial: a Survey on Diagnosis and Prevention of Catheter-Related Infections in Patients on Home Parenteral Nutrition
Brief Title: The AOT (Acridine Orange and Taurolidine) Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: G.Wanten, MD, PhD, MSc, Dept of Gastroenterology and Hepatology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AOT-trial
Record Dates: First submitted 2006-05-02; First posted 2006-05-03 (Estimated); Last update posted 2009-02-11 (Estimated); Status verified 2009-02

CONDITIONS: Parenteral Nutrition; Infection; Sepsis
Keywords: nutrition; parenteral; infection; katheter; taurolidine; acridine orange; prevention
MeSH Terms: conditions — Hyperphagia; Infections; Sepsis | interventions — taurolidine

INTERVENTIONS:
Drug: taurolidine

SUMMARY:
Total parenteral (intravenous) nutrition in the home setting (Home TPN or HPN) is a life saving strategy in patients who suffer from severe intestinal failure. Unfortunately, this treatment modality remains complicated by the development of frequent infectious complications. This especially relates to the device that is used to establish venous access, mostly a catheter (Hickman-Broviac type) or a port-a-cath.

Taurolodine is an antimicrobial agent without any known side effects or resistance-related problems that holds promise as an effective antibiotic lock solution to prevent catheter infections, as demonstrated recently in a pilot study in HPN patients [Jurewitsch, 2005].

In addition, recently a test has been described which may enable to confirm a suspected diagnosis of central line infection within one hour, the so-called Acridine Orange Leukocyte Cytospin test (AOLC) [Bong, 2003]. For this test, blood that is drawn from the central line is stained with the fluorescent dye acridine orange. Next, microscopic evaluation for the presence of micro-organisms takes place. Implementation of this test might enable to start treatment of the infection and prevent unnecessary removal of non-infected central lines without the necessity to several days wait for culture results.

DETAILED DESCRIPTION:
Two hypotheses will be tested in the AOT trial:

1. The use of taurolidine as an antibiotic lock (5 mL) to flush the central line after infusing the TPN formulation, when compared to the present use of heparin solution (5 mL, 150 E/mL) decreases the rate of catheter-related infections in HPN patients
2. Implementation of the acridine orange staining test allows an earlier diagnosis (or rejection of this diagnosis) compared to culture results. Importantly, in the present trial the results of this test will not be used for treatment decisions.

To this end, patients who are admitted to the clinical ward because of suspected central line infection (mostly because of fever and/or chills) will be treated according to the current protocol for catheter sepsis, after obtaining central line and peripheral blood cultures. This protocol includes the administration of medicinase through the central line and i.v. antibiotics peripherally. After obtaining informed consent, in addition 5 cc of EDTA blood will be drawn from the central line to perform (within 24 hours) the acridine orange cytospin staining test and a Gram stain. These results will than be compared to the culture results. Based on culture results, the antibiotics will be tailored.

If the patient recovers and TPN administration can be restarted, randomisation between heparin lock (5 mL, 150 E/mL) versus taurolidine lock solution 2% (5 mL) will take place. In case the catheter has to be removed because of ongoing or recurrent sepsis, randomisation takes place after a new central line has been placed and the patient continues on TPN.

A new episode of proven catheter sepsis is considered as the primary end-point.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* patient on home TPN with central line (Hickman or Porth-a-cath)
* suspected central line infection (acridine orange test)
* proven central line infection (randomisation tauroline vs heparin)

Exclusion Criteria:

* no informed consent
* patient on home TPN with arteriovenous fistula (shunt)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-06; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
time between episodes of central line infection in one patient

SECONDARY OUTCOMES:
outcome of acridine orange staining test compared to culture results

CONTACTS AND LOCATIONS:
Overall Officials: Geert Wanten, MD, PhD, Principal Investigator — Radboud University Nijmegen Medical Centre, The Netherlands
Locations (1):
- Department of Gastroenterology and Hepatology clinical ward, Nijmegen, Netherlands

REFERENCES:
- [Background] Jurewitsch B, Jeejeebhoy KN. Taurolidine lock: the key to prevention of recurrent catheter-related bloodstream infections. Clin Nutr. 2005 Jun;24(3):462-5. doi: 10.1016/j.clnu.2005.02.001. Epub 2005 Apr 22. PMID 15896434
- [Background] Bong JJ, Kite P, Ammori BJ, Wilcox MH, McMahon MJ. The use of a rapid in situ test in the detection of central venous catheter-related bloodstream infection: a prospective study. JPEN J Parenter Enteral Nutr. 2003 Mar-Apr;27(2):146-50. doi: 10.1177/0148607103027002146. PMID 12665171
- [Derived] Bisseling TM, Willems MC, Versleijen MW, Hendriks JC, Vissers RK, Wanten GJ. Taurolidine lock is highly effective in preventing catheter-related bloodstream infections in patients on home parenteral nutrition: a heparin-controlled prospective trial. Clin Nutr. 2010 Aug;29(4):464-8. doi: 10.1016/j.clnu.2009.12.005. Epub 2010 Jan 12. PMID 20061070